CLINICAL TRIAL: NCT02599584
Title: Improvement of Team Performance With a Pre-critical Staff Within the Team Prior to Admission of Critical Simulated Patient in High Fidelity Simulation Session for Anesthesiology Resident During Their Education Curriculum
Brief Title: Performance and Team Pre-critical Staff Before Critical Event in High Fidelity Simulation for Anesthesiology Residents
Acronym: Simstaf&perf
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Claude Bernard University (Other)
Responsible Party: Principal Investigator, Lilot Marc, MD, Claude Bernard University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: CLESS 2015
Record Dates: First submitted 2015-11-04; First posted 2015-11-06 (Estimated); Last update posted 2020-03-02 (Actual); Status verified 2020-02

CONDITIONS: Healthy
Keywords: behaviour
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- precritical staff (Experimental): 4 min of precritical team staff for anticipation of risk and role attribution during the critical events if they occur. athe staff will take place after briefing of the scenario and before the start of the scenario.
  Interventions: Behavioral: precritical staff
- control (No Intervention): screening of normal labs results during 4 min, after briefing of the scenario and before the start of the scenario

INTERVENTIONS:
Behavioral: precritical staff — free pre critical scenario team staff
  Arms: precritical staff

SUMMARY:
Simulated environment allowed safe learning of critical events and knowledge of appropriate response and treatment. Anesthesiology resident education curriculum in Lyon plans several high fidelity simulation session with a large panel of critical events. Anticipation of critical events before they may occur and plannification of team resources and priority in the treatment strategy may help to improve team performance during the scenario. The investigators' goal is to compare team performance during the scenario with or without a liberal preparation team staff of 4 min, suggested after the briefing of the scenario but before the scenario starts.

DETAILED DESCRIPTION:
High fidelity simulated environment allowed safe learning of critical events and knowledge of appropriate response and treatment. Anesthesiology resident education curriculum in Lyon plans several high fidelity simulation session with a large panel of critical events. Anticipation of critical events before they may occur, plannification of team resources, priority in the treatment strategy and effective communication within the team, may help to improve team performance during the scenario. The investigators' goal is to compare team performance during the scenario with or without a preparation team staff of 4 min. This staff will be suggested after the briefing of the scenario but before the scenario starts. The investigators are going to compare groups of anesthesiology residents going through same scenarios of simulated critical events in high fidelity simulation session. Scenarios will be recorded to be analyzed by 2 reviewers independantly. A checklist of appropriate treatment and a non technical skill checklist will be use to cote team performance. Stress of the participants will be assessed by visual analogic scale of participants anxiety and stress. the two groups (preparation staff or no preparation staff) will be compare to see if improvement in team performance is associated with the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Anesthesiology resident in the education simulation curriculum

Exclusion Criteria:

* no verbal consent

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2015-11; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
performance | one week (review video)
  performance scale cotation (rated from 0 to 100 by 2 independant experts) (technikal and non technikal skills scale)

SECONDARY OUTCOMES:
stress | min 0, min 4 and min 15 (just after the scenario)
  visual analogic scale (transfer to metrics from 0 to 100) of the stress felt by the residents at the time of the cotation

CONTACTS AND LOCATIONS:
Overall Officials: jean jacques lehot, PHD, Study Chair — CLESS
Locations (1):
- CLESS, Lyon, Auvergne-Rhône-Alpes, France

IPD SHARING:
Plan to Share IPD: Undecided